CLINICAL TRIAL: NCT06652984
Title: Effectiveness of Respiratory Muscle Training Using a Mobile Respiratory Trainer in People With Ankylosing Spondylitis
Brief Title: Effectiveness of Mobile Respiratory Training in Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ayk-AirPro; 119-2024/SB002 (Other: Usak University Scientific Research Projects)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Ankylosing Spondylitis; Respiratory Distress; Exercise Therapy; Breath Tests
Keywords: rheumatological diseases; respiratory exercises; Lung capacity
MeSH Terms: conditions — Spondylitis, Ankylosing; Dyspnea

STUDY DESIGN:
Intervention Model Description: Randomized pretest-posttest parallel group design
Who Masked: Outcomes Assessor
Masking Description: A blind physiotherapist will be in charge of the assessment of the outcomes of the study in all patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercisers with a mobile breathing apparatus (Active Comparator): The mobile device will be given to the patient for use. The exercise programme will be taught by the physiotherapist with face-to-face training before the study. The settings of the device will be started at the beginner level in breathing and exhalation exercises.
  Interventions: Other: Exercise 1
- Pursed Lip Breathing Exercisers (Active Comparator): 'Pursed lip breathing' will be taught to the patients in this group. The programme will be taught by the physiotherapist with face-to-face training before the study. The patient will be taught to take a deep breath through the nose as much as he/she can and then to empty the air in the lungs in a controlled manner without applying any force by pursing the lips as if whistling.
  Interventions: Other: Exercise 2

INTERVENTIONS:
Other: Exercise 1 — Patients were planned to complete exercise sessions 5 times a week for 12 weeks, each lasting 35 minutes per day.
  Arms: Exercisers with a mobile breathing apparatus
Other: Exercise 2 — Patients were planned to complete exercise sessions 5 times a week for 12 weeks, each lasting 35 minutes per day.
  Arms: Pursed Lip Breathing Exercisers

SUMMARY:
Introduction and aim; Low functionality of respiratory muscles is frequently observed in various diseases such as chronic obstructive pulmonary disease, cystic fibrosis, idiopathic pulmonary fibrosis, and rheumatological diseases such as ankylosing spondylitis. Strengthening the respiratory muscles is a part of the treatment in such disease groups, and it has been reported that the quality of life of patients increases with the improvement in the respiratory muscles. Stavrou et al. In a study published in 2021, they achieved an increase in VO2max and maximum respiratory power in athletes after an exercise program with the AirOFit PRO™ (AirOFit, Copenhagen, Denmark) branded mobile breathing exercise device, which they introduced as a new technology. However, there is no study yet reporting the use of this device in rheumatological diseases.

The aim of this study is to investigate the effects of personalized breathing exercises with the AirOFit PRO™ (AirOFit, Copenhagen, Denmark) branded mobile breathing exercise device on respiratory muscles and functional exercise capacity, as well as on specific outcomes of the disease, in patients with ankylosing spondylitis.

Hypotheses of the study;

a) Hypothesis H1: Personalised breathing exercises applied with a mobile respiratory exercise device in patients with ankylosing spondylitis have a positive effect on respiratory capacity and activities of daily living in patients.

DETAILED DESCRIPTION:
Inflammation of the thoracic and costovertebral joints in ankylosing spondylitis causes gradual fusion and ossification over time, which adversely affects costal mobility and thoracic expansion. In some patients, this leads to increased dorsal kyphosis, thoracic stiffness and permanent limitation of chest wall motion. Expansion and reduced lung volume as a result of mechanical constriction caused by ankylosis of the thoracic joints explains the restrictive breathing pattern in these patients. In addition, previous studies have shown that the inflammatory process of the disease causes pain and stiffness in the thoracic joints, contributing to decreased respiratory function. It is thought that breathing exercises that strengthen the inspiratory muscles may prevent or delay complications that may occur due to inspiratory muscle weakness. Previous studies in the literature have examined the effectiveness of inspiratory muscle training in different disease groups. However, few studies in patients with ankylosing spondylitis have examined the effect of inspiratory muscle training on pulmonary function and aerobic capacity. According to our current knowledge, there is no academic study in the international literature using the mobile respiratory exercise device AirOFit PRO™ (AirOFit, Copenhagen, Denmark) for personalised respiratory exercise in any rheumatic disease.

According to our current knowledge, there is no academic study in the international literature using the AirOFit PRO™ (AirOFit, Copenhagen, Denmark) mobile respiratory exercise device for personalised respiratory exercise in any rheumatic disease. This study will be the first study to evaluate the effectiveness of a daily sustainable respiratory exercise programme suitable for home use in rheumatic patients and will be included in the international literature. In addition, it will be the basis for academic studies that enable long-term follow-up of patients with this mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer for the study
* Be over 18 years old
* To be in the follow-up of Usak University Rheumatology outpatient clinic
* Stability in medical treatment (keeping disease activity under control with the same medical treatment for at least 6 months)

Exclusion Criteria:

* The presence of diseases that affect the function of the respiratory system (such as pneumonia, pleurisy, empyema, pneumothorax, hemothorax, hydrothorax, atelectasis, pulmonary oedema, pulmonary hypertension, emphysema, and lung cancer).
* The presence of a regular exercise habit (regularly 3 days a week for at least six months).
* Significant physical disability or impairment (regular use of walking aids, etc.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Tidal volume | At the end of the 12th week of exercise schedule
  Tidal volume; This is the amount of air breathed in or out during normal breathing. This pulmonary function test will done with a spirometry.
Vital capacity | At the end of the 12th week of exercise schedule
  This is the total volume of air that can be breathed out after breathing in as much as you can. This pulmonary function test will done with a spirometry.
Forced vital capacity | At the end of the 12th week of exercise schedule
  Forced vital capacity (FVC); This is the amount of air breathed out forcefully and quickly after breathing in as much as you can. This pulmonary function test will done with a spirometry.

SECONDARY OUTCOMES:
The Bath Ankylosing Spondylitis Functional Index | At the end of the 12th week of exercise schedule
  The Bath Ankylosing Spondylitis Functional Index (BASFI) is a set of 10 questions designed to determine the degree of functional limitation in patients with Ankylosing Spondylitis (AS). The 10 questions were chosen with a major input from patients with AS. The first 8 questions are about everyday tasks and dependent on functional anatomy (bending, reaching, changing position, standing, turning, and climbing steps with or without rail) while the final 2 questions assess the patients' ability to cope with everyday life. Each item is scored on a scale of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y KARAHAN, MD, Principal Investigator — Uşak University
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing personal data must comply with the data protection principles in Turkey.

REFERENCES:
- [Result] Stavrou VT, Tourlakopoulos KN, Daniil Z, Gourgoulianis KI. Respiratory Muscle Strength: New Technology for Easy Assessment. Cureus. 2021 May 2;13(5):e14803. doi: 10.7759/cureus.14803. PMID 34094759